CLINICAL TRIAL: NCT04695015
Title: Research of Pathological Imaging Diagnosis of Ocular Tumors Based on New Artificial Intelligence Algorithm
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Chun Zhang, professor, Peking University
Other Study IDs: IRB00006761-M2020434
Record Dates: First submitted 2020-11-19; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Melanoma (Skin); Melanoma in Situ; Nevus Eye; Sebaceous Gland Carcinoma of the Eyelid; Basal Cell Carcinoma; Squamous Cell Carcinoma in Situ; Ocular Tumor
MeSH Terms: conditions — Melanoma; Carcinoma, Basal Cell; Squamous Intraepithelial Lesions; Eye Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — After the blood samples are treated with EDTA anti coagulation, the second-generation sequencing is performed from the DNA level and the RNA level to collect relevant genomics information, and establish an ocular tumor fusion genome database. Investigators will establish a complete sequencing data annotation database based on the existing tumor sequencing data annotation and analysis of soft nail sets and tumor sequencing data related public databases (such as the cosmic database).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Melanoma and Nevus: Patients diagnosed with melanoma or/and nevus on the skin around the eye before surgery.
- Basal cell carcinoma;Squamous cell carcinoma;Sebaceous gland carcinoma: Patients diagnosed with basal cell carcinoma, squamous cell carcinoma, sebaceous gland carcinoma before surgery.

SUMMARY:
The purpose of this study is to establish a standardized process for obtaining digital pathological image information of ocular tumors; use modern pathological techniques to obtain the co-expression information of multiple biomarkers in the pathological tissues of ocular tumors, and finally construct standardized digital ocular tumors with biomarkers Pathology image database.

DETAILED DESCRIPTION:
This study is a prospective study. Patients with common and representative ocular tumors in the Department of Ophthalmology, Peking University Third Hospital, will be selected and enrolled after informed consent to collect basic clinical information, preoperative blood samples, and ocular tumors Obtain pathological image annotation data and genomics-related data from ocular tumor tissue specimens, use blood samples for genomics information analysis, provide multi-dimensional data for the development of artificial intelligence algorithms, and establish artificial intelligence-assisted image data for eye tumors Standardize the process and establish a multi-modal ocular tumor standardized database of "clinical information-tissue samples-pathological images-genomics data". The database and the diagnosis system are correlated with each other to provide optimal image data for later machine learning and related algorithm establishment, and finally the investigators will be completed the design of a new artificial intelligence-assisted diagnosis system for eye tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with eye tumors and undergoing eye tumor surgery.
2. Patients sign informed consent for sample collection and sample transfer agreement, and can cooperate with long-term regular follow-up requirements.

Exclusion Criteria:

1. Patients who are unable to undergo tumor surgery or retain samples due to various reasons .
2. Patients who are positive for hepatitis B, HIV, and syphilis.
3. Patient compliance is poor.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients from the Department of Ophthalmology, Peking University Third Hospital who has an eye tumor and undergoes surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-31 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
To compare the diagnostic accuracy of OPAL and IHC for melanoma and other tumors. | Up to 24 weeks.
  The result of OPAL automatic analysis will be compared with IHC manual counting analysis.The accuracy of the study will be declared "success" if OPAL automatic analysis meet more than 85% of the manual count for all antibody.

CONTACTS AND LOCATIONS:
Overall Officials: Chun Zhang, MD/PHD, Principal Investigator — Peking University Third Hospital